CLINICAL TRIAL: NCT00559897
Title: Phase II Study Evaluating the Effect of Zolendronic Acid on Standardized Uptake Value (SUV) on FLT PET Scans in Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Zoledronic Acid and Positron Emission Tomography in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shirish Gadgeel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000543463; P30CA022453 (NIH); WSU-2006-136 (Other: Karmanos Cancer Institute)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: bone metastases; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3'-deoxy-3'-[18F]FLT PET & zoledronic acid (Experimental): Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid
  Single photon emission computed tomography. Patient should receive the dose of zoledronic acid within 48 hrs of the first '3'-deoxy-3'-[18F]FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.
  Interventions: Other: 3'-deoxy-3'-[18F]FLT; Procedure: Single photon emission computed tomography

INTERVENTIONS:
Other: 3'-deoxy-3'-[18F]FLT — Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.
Procedure: Single photon emission computed tomography — Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.

SUMMARY:
RATIONALE: A positron emission tomography scan is a procedure in which a small amount of radioactive sugar is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where tumor cells are found. This study is looking at whether the drug zoledronic acid interferes with the ability of a PET scan to find tumor cells.

PURPOSE: This phase II trial is studying how well positron emission tomography works when given together with zoledronic acid in finding tumor cells in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the PET response rate after zoledronic acid in patients with non-small cell lung cancer.

OUTLINE: Patients receive 1 dose of zoledronic acid on day 1 followed by 3'-deoxy-3'-[18F]fluorothymidine/PET to determine standardized uptake value.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB (with pleural effusion) or stage IV disease
* Candidate for systemic therapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No active brain metastases

  * More than 7 days since prior radiotherapy for brain metastases
  * Must be neurologically stable with no seizures within the past 3 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN (5 times ULN if liver metastases present)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min by Cockcroft-Gault formula
* No current active dental problems, including infection of the teeth or jawbone (maxilla or mandible)
* No dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw, of exposed bone in the mouth, or of slow healing after dental procedures
* Not pregnant
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior or other concurrent bisphosphonates
* More than 2 weeks since prior surgery
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 7 days since prior palliative radiotherapy and recovered
* More than 6 weeks since prior and no planned dental or jaw surgery
* More than 30 days since prior participation in an investigational trial
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid: Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid
  Single photon emission computed tomography. Patient should receive the dose of zoledronic acid within 48 hrs of the first '3'-deoxy-3'-[18F]FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.
  3'-deoxy-3'-[18F]FLT: Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.
  Single photon emission computed tomography: Patient should receive the dose of zoledronic acid within 48 hours of the first FLT PET scan. The second FLT PET scan will be done 6-8 days after the dose of zoledronic acid.
Period: Overall Study
Arm/Group | 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: PET Response Rate
Time Frame: FLT PET scan will be done 6-8 days after the dose of zoledronic acid
Arm/Group | 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At week 3
Arm/Group | 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3'-Deoxy-3'-[18F]FLT PET & Zoledronic Acid (N=6)
Altered Mental Status (Psychiatric disorders) | 1 (1) — Related to brain mets

LIMITATIONS AND CAVEATS:
None of the participants were evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes